CLINICAL TRIAL: NCT04217876
Title: Clinical, Morphological and Functional Aspects in Acute and Chronic Myocarditis.
Brief Title: Clinical, Morphological and Functional Aspects in Myocarditis.
Status: Completed | Type: Observational
Sponsor: University of Messina (Other)
Collaborators: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government); Humanitas Hospital, Italy (Other); Vannini Hospital Rome (Unknown)
Responsible Party: Principal Investigator, Gianluca Di Bella, Associate Professor Cardiovascular Diseases, University of Messina
Other Study IDs: 11616
Record Dates: First submitted 2019-12-28; First posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Myocarditis
Keywords: echocardiography; cardiac magnetic resonance; myocarditis
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinically suspected infarct-like acute myocarditis: Diagnosis of infarct-like AM was based on five criteria: (a) history of flu-like symptoms within 8 weeks prior admission; (b) new onset of symptoms such as fatigue/breathlessness, chest pain, mild dyspnea, and/or palpitation; (c) ischemic ECG pattern (ST-segment elevation and/or T-wave anomalies); (d) increase of inflammatory markers (non-high- sensitivity CRP > 8 mg/L and/or white blood cell count > 11.000/mm3) and cardiac enzymes; and (e) preserved global systolic function (EF > 50%). We excluded patients with New York Heart Association (NYHA) functional heart classifications II-IV, LVEF < 50% and those patients with electrocardiographic evidence of bradyarrhythmias (≥second-degree atrioventricular block) or tachyarrhythmias (ventricular or supraventricular arrhythmias).
  Interventions: Diagnostic Test: post-processing analysis of cardiac imaging (strain echocardiography)

INTERVENTIONS:
Diagnostic Test: post-processing analysis of cardiac imaging (strain echocardiography) — A dedicated software package for two-dimensional speckle tracking strain analysis (XStrain™, Esaote, Florence, Italy) was used to quantify both ENDO and EPI strains. Our echocardiographic imaging acquisition protocol for 2DSTE consisted in the acquisition of three consecutive cardiac cycles from non-foreshortened apical views (4, 2, and 3 chambers) obtained during breath hold. Frame-by- frame displacement of ENDO and EPI points was automatically evaluated, generating strain curves for each segment.
  The tracking quality was verified for each segment, and subsequent manual adjustments were performed, when required. All data were analyzed with the aid of Fourier techniques, which ensure greater accuracy using the periodicity of the heart motion.

SUMMARY:
Cardiac magnetic resonance (CMR) is accurate to identify acute myocardial damage (edema, hyperemia, and/or fibrosis) due to acute myocarditis (AM). Recently, two-dimensional strain echocardiography was also validated in order to provide important information on myocardial dysfunction in patients with AM, even if no wall motion abnormalities are detected. No data are available about incidence of longitudinal myocardial dysfunction and its prognostic role in AM.

DETAILED DESCRIPTION:
In this study, the investigators will analyze the effect of acute myocarditis-induced damage on LV myocardial deformation and remodeling both in the acute myocarditis phase and follow-up period (about 2 years later). The investigators will use a combined approach including strain echocardiography to asses left ventricular myocardial deformation and late gadolinium enhancement (LGE)cardiac magnetic resonance for the assessment of left ventricular damage.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of clinical suspected acute myocarditis (AM)
* diagnosis of AM with cardiac magnetic resonance (CMR) according to Lake Louise criteria (myocardial edema, hyperemia, and LGE).
* absence of coronary artery diseases confirmed by coronary angiography or computed tomography in all patients with the exception of those younger than 30 years with a low risk of coronary artery disease.

Exclusion Criteria:

* Previous heart diseases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive in-patients with a definite CMR diagnosis of AM having a follow-up CMR examination including cine CMR, T1, T2 weighted and LGE images.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Demonstrating incidence of longitudinal dysfunction of left ventricle in patients with acute myocarditis and preserved ejection fraction. | Day 0
  Longitudinal systolic function (s-1) of the left ventricle will be measured (%) by echocardiography.
Demonstrating effect of myocarditis damage due to myocardial fibrosis on longitudinal function. | Day 0
  Longitudinal systolic function (s-1) of the left ventricle will be measured (%) by echocardiography.
  Myocardial fibrosis LGE was defined as myocardium with an signal intensity higher than the average signal intensity of the region of interest more than 6 standard deviation in late gadolinium enhancement technique.

SECONDARY OUTCOMES:
Prognostic role of longitudinal dyfunction. | from 6-60 months
  cardiac death, resuscitated cardiac arrest, ventricular assist device implantation, cardiac transplantation, appropriate implantable cardioverter defibrillator (ICD) shock, relapse of AM and hospitalization for worsening heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Di Bella, Principal Investigator — University of Messina, Italy; Mariapaola Campisi, MD, Study Chair — University of Messina, Italy
Locations (4):
- Italy (4):
  - Lorenzo Monti, Milan
  - Alessandro Pingitore, Pisa
  - Giovanni D Aquaro, Pisa
  - Giovanni Camastra, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aretz HT, Billingham ME, Edwards WD, Factor SM, Fallon JT, Fenoglio JJ Jr, Olsen EG, Schoen FJ. Myocarditis. A histopathologic definition and classification. Am J Cardiovasc Pathol. 1987 Jan;1(1):3-14. No abstract available. PMID 3455232
- [Result] Leone O, Veinot JP, Angelini A, Baandrup UT, Basso C, Berry G, Bruneval P, Burke M, Butany J, Calabrese F, d'Amati G, Edwards WD, Fallon JT, Fishbein MC, Gallagher PJ, Halushka MK, McManus B, Pucci A, Rodriguez ER, Saffitz JE, Sheppard MN, Steenbergen C, Stone JR, Tan C, Thiene G, van der Wal AC, Winters GL. 2011 consensus statement on endomyocardial biopsy from the Association for European Cardiovascular Pathology and the Society for Cardiovascular Pathology. Cardiovasc Pathol. 2012 Jul-Aug;21(4):245-74. doi: 10.1016/j.carpath.2011.10.001. Epub 2011 Dec 3. PMID 22137237
- [Result] Caforio AL, Pankuweit S, Arbustini E, Basso C, Gimeno-Blanes J, Felix SB, Fu M, Helio T, Heymans S, Jahns R, Klingel K, Linhart A, Maisch B, McKenna W, Mogensen J, Pinto YM, Ristic A, Schultheiss HP, Seggewiss H, Tavazzi L, Thiene G, Yilmaz A, Charron P, Elliott PM; European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Current state of knowledge on aetiology, diagnosis, management, and therapy of myocarditis: a position statement of the European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Eur Heart J. 2013 Sep;34(33):2636-48, 2648a-2648d. doi: 10.1093/eurheartj/eht210. Epub 2013 Jul 3. PMID 23824828
- [Result] Belkaya S, Kontorovich AR, Byun M, Mulero-Navarro S, Bajolle F, Cobat A, Josowitz R, Itan Y, Quint R, Lorenzo L, Boucherit S, Stoven C, Di Filippo S, Abel L, Zhang SY, Bonnet D, Gelb BD, Casanova JL. Autosomal Recessive Cardiomyopathy Presenting as Acute Myocarditis. J Am Coll Cardiol. 2017 Apr 4;69(13):1653-1665. doi: 10.1016/j.jacc.2017.01.043. PMID 28359509
- [Result] Friedrich MG, Sechtem U, Schulz-Menger J, Holmvang G, Alakija P, Cooper LT, White JA, Abdel-Aty H, Gutberlet M, Prasad S, Aletras A, Laissy JP, Paterson I, Filipchuk NG, Kumar A, Pauschinger M, Liu P; International Consensus Group on Cardiovascular Magnetic Resonance in Myocarditis. Cardiovascular magnetic resonance in myocarditis: A JACC White Paper. J Am Coll Cardiol. 2009 Apr 28;53(17):1475-87. doi: 10.1016/j.jacc.2009.02.007. PMID 19389557
- [Result] Aquaro GD, Ghebru Habtemicael Y, Camastra G, Monti L, Dellegrottaglie S, Moro C, Lanzillo C, Scatteia A, Di Roma M, Pontone G, Perazzolo Marra M, Barison A, Di Bella G; "Cardiac Magnetic Resonance" Working Group of the Italian Society of Cardiology. Prognostic Value of Repeating Cardiac Magnetic Resonance in Patients With Acute Myocarditis. J Am Coll Cardiol. 2019 Nov 19;74(20):2439-2448. doi: 10.1016/j.jacc.2019.08.1061. PMID 31727281
- [Result] Aquaro GD, Camastra G, Monti L, Lombardi M, Pepe A, Castelletti S, Maestrini V, Todiere G, Masci P, di Giovine G, Barison A, Dellegrottaglie S, Perazzolo Marra M, Pontone G, Di Bella G; working group "Applicazioni della Risonanza Magnetica" of the Italian Society of Cardiology. Reference values of cardiac volumes, dimensions, and new functional parameters by MR: A multicenter, multivendor study. J Magn Reson Imaging. 2017 Apr;45(4):1055-1067. doi: 10.1002/jmri.25450. Epub 2016 Aug 29. PMID 27571232
- [Result] Aquaro GD, Perfetti M, Camastra G, Monti L, Dellegrottaglie S, Moro C, Pepe A, Todiere G, Lanzillo C, Scatteia A, Di Roma M, Pontone G, Perazzolo Marra M, Barison A, Di Bella G; Cardiac Magnetic Resonance Working Group of the Italian Society of Cardiology. Cardiac MR With Late Gadolinium Enhancement in Acute Myocarditis With Preserved Systolic Function: ITAMY Study. J Am Coll Cardiol. 2017 Oct 17;70(16):1977-1987. doi: 10.1016/j.jacc.2017.08.044. PMID 29025554
- [Result] Aquaro GD, Negri F, De Luca A, Todiere G, Bianco F, Barison A, Camastra G, Monti L, Dellegrottaglie S, Moro C, Lanzillo C, Scatteia A, Di Roma M, Pontone G, Perazzolo Marra M, Di Bella G, Donato R, Grigoratos C, Emdin M, Sinagra G. Role of right ventricular involvement in acute myocarditis, assessed by cardiac magnetic resonance. Int J Cardiol. 2018 Nov 15;271:359-365. doi: 10.1016/j.ijcard.2018.04.087. Epub 2018 Jul 22. PMID 30045820
- [Result] Lopez-Ayala JM, Pastor-Quirante F, Gonzalez-Carrillo J, Lopez-Cuenca D, Sanchez-Munoz JJ, Oliva-Sandoval MJ, Gimeno JR. Genetics of myocarditis in arrhythmogenic right ventricular dysplasia. Heart Rhythm. 2015 Apr;12(4):766-73. doi: 10.1016/j.hrthm.2015.01.001. Epub 2015 Jan 20. PMID 25616123
- [Result] Di Bella G, Minutoli F, Pingitore A, Zito C, Mazzeo A, Aquaro GD, Di Leo R, Recupero A, Stancanelli C, Baldari S, Vita G, Carerj S. Endocardial and epicardial deformations in cardiac amyloidosis and hypertrophic cardiomyopathy. Circ J. 2011;75(5):1200-8. doi: 10.1253/circj.cj-10-0844. Epub 2011 Mar 17. PMID 21427499